CLINICAL TRIAL: NCT01602692
Title: A Comparison of Tumescence in Breast Reduction Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-0543; A539730 (Other: UW, Madison); SMPH/SURGERY/DENT&P SRG (Other: UW, Madison)
Record Dates: First submitted 2012-05-04; First posted 2012-05-21 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: Pain, postoperative; Postoperative Nausea and Vomiting; Patient Readmission; Time to Discharge
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tumescent solution with dilute epinephrine (Active Comparator): Subjects in this arm of the study will be randomized to receive tumescent solution containing dilute epinephrine (1:1,000,000) during their breast reduction.
  Interventions: Drug: Tumescent Solution with dilute epinephrine
- Tumescent solution with dilute lidocaine and epinephrine (Active Comparator): Subjects in this arm of the study will receive tumescent solution containing both dilute lidocaine (0.05%) and dilute epinephrine (1:1,000,000).
  Interventions: Drug: Tumescent solution with dilute lidocaine and epinephrine

INTERVENTIONS:
Drug: Tumescent solution with dilute lidocaine and epinephrine — Tumescent Solution containing both dilute lidocaine (0.05%) and dilute epinephrine (1:1,000,000)
  Arms: Tumescent solution with dilute lidocaine and epinephrine
Drug: Tumescent Solution with dilute epinephrine — Tumescent Solution containing dilute epinephrine (1:1,000,000) only
  Arms: Tumescent solution with dilute epinephrine

SUMMARY:
The investigators' main hypothesis is that in breast reduction surgery, the use of tumescent solution containing both dilute lidocaine and epinephrine will lead to better control of postoperative pain, nausea, vomiting, shorter time through postoperative phases of care, quicker discharge from the hospital and lower numbers of hospital readmissions than the use of tumescent solution containing only dilute epinephrine.

DETAILED DESCRIPTION:
Postoperative pain is often undermanaged in surgical patients. In the outpatient surgery population, such as breast reduction surgery, postoperative pain can lead to increased narcotic use, increased nausea, surgical complications and unplanned hospital admission, in addition to patient discomfort or dissatisfaction. Tumescence is a method of infiltrating tissues, such as the breast, with solutions of very dilute lidocaine and/or very dilute epinephrine in order to provide diffuse local anesthesia, hemostasis, and tissue manipulation. Both types of solution are considered standard care and both at the University of Wisconsin, Madison. There are two main aims to this study. Aim 1 is to determine the effect of dilute lidocaine in tumescent solution on post-operative pain following breast reduction surgery. Aim 2 of our study is to determine the effect of dilute lidocaine in tumescent solution on secondary post-operative outcomes following breast reduction surgery. The secondary outcomes that will be measured in this study include average time (minutes) spent in the postanesthesia care unit (PACU), average time (minutes) spent in Phase 2, total time (minutes) between the end of case and discharge home, occurrence of unplanned hospital admission, number of episodes of post-operative nausea (subjective feeling vs. emesis) and amount of anti-emetic medication used in pacu, phase 2 and the first 24 hours post-op (mg). The investigators hypothesize that tumescence with lidocaine and epinephrine will have improved post-operative pain control leading to less narcotic use during the first twenty four hours postoperatively. (Aim 1). The investigators also believe that tumescence with lidocaine and epinephrine will lead to less time spent in PACU, less time spent in Phase2, less time between the end of the case and discharge home, less occurrence of unplanned hospital admissions, less episodes of post-operative nausea and less amount of antiemetic medication used in PACU, phase 2 and the first 24 hours post-op (Aim 2). The investigators propose that such differences could play a significant role in surgical outcomes and patient satisfaction in outpatient plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting for breast reduction surgery at the University of Wisconsin Hospital and Clinics and the University of Wisconsin Transformations Surgery Center and who do not meet any of the exclusion criteria.

Exclusion Criteria:

* Women under the age of 18 years
* Breast feeding or pregnant women
* Incarcerated women.
* Women unable to give consent because of impaired decision making ability.
* Women who have reported allergies to the substances that will be used in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkat K Rao, M.D. M.B.A, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Transformations Surgery Center, Middleton, Wisconsin, United States

REFERENCES:
- [Background] Lu L, Fine NA. The efficacy of continuous local anesthetic infiltration in breast surgery: reduction mammaplasty and reconstruction. Plast Reconstr Surg. 2005 Jun;115(7):1927-34; discussion 1935-6. doi: 10.1097/01.prs.0000163332.04220.bd. PMID 15923838
- [Background] Rawlani V, Kryger ZB, Lu L, Fine NA. A local anesthetic pump reduces postoperative pain and narcotic and antiemetic use in breast reconstruction surgery: a randomized controlled trial. Plast Reconstr Surg. 2008 Jul;122(1):39-52. doi: 10.1097/PRS.0b013e3181774349. PMID 18594373
- [Background] Kryger ZB, Rawlani V, Lu L, Fine NA. Decreased postoperative pain, narcotic, and antiemetic use after breast reduction using a local anesthetic pain pump. Ann Plast Surg. 2008 Aug;61(2):147-52. doi: 10.1097/SAP.0b013e31815a23ef. PMID 18650606
- [Background] Schurr MJ, Gordon DB, Pellino TA, Scanlon TA. Continuous local anesthetic infusion for pain management after outpatient inguinal herniorrhaphy. Surgery. 2004 Oct;136(4):761-9. doi: 10.1016/j.surg.2004.06.016. PMID 15467660
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Quality improvement guidelines for the treatment of acute pain and cancer pain. American Pain Society Quality of Care Committee. JAMA. 1995 Dec 20;274(23):1874-80. doi: 10.1001/jama.1995.03530230060032. PMID 7500539
- [Background] Klein JA. Tumescent technique for regional anesthesia permits lidocaine doses of 35 mg/kg for liposuction. J Dermatol Surg Oncol. 1990 Mar;16(3):248-63. doi: 10.1111/j.1524-4725.1990.tb03961.x. PMID 2179348
- [Background] Ostad A, Kageyama N, Moy RL. Tumescent anesthesia with a lidocaine dose of 55 mg/kg is safe for liposuction. Dermatol Surg. 1996 Nov;22(11):921-7. doi: 10.1111/j.1524-4725.1996.tb00634.x. PMID 9063507
- [Background] Larson JD, Gutowski KA, Marcus BC, Rao VK, Avery PG, Stacey DH, Yang RZ. The effect of electroacustimulation on postoperative nausea, vomiting, and pain in outpatient plastic surgery patients: a prospective, randomized, blinded, clinical trial. Plast Reconstr Surg. 2010 Mar;125(3):989-94. doi: 10.1097/PRS.0b013e3181ccdc23. PMID 20195124
- [Background] Heller L, Kowalski AM, Wei C, Butler CE. Prospective, randomized, double-blind trial of local anesthetic infusion and intravenous narcotic patient-controlled anesthesia pump for pain management after free TRAM flap breast reconstruction. Plast Reconstr Surg. 2008 Oct;122(4):1010-1018. doi: 10.1097/PRS.0b013e3181858c09. PMID 18827631
- [Result] Christie BM, Kapur S, Kempton SJ, Hanson SE, Ma Y, Rao VK. A Prospective Randomized Trial Comparing the Effects of Lidocaine in Breast Reduction Surgery. Plast Reconstr Surg. 2017 May;139(5):1074e-1079e. doi: 10.1097/PRS.0000000000003243. PMID 28445354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: female candidates presenting for bilateral breast reduction at the University of Wisconsin ambulatory surgery center performed by a single surgeon (Dr. Rao)
Groups:
- Tumescent Solution With Dilute Epinephrine: Participants in this arm of the study will be randomized to receive tumescent solution containing dilute epinephrine (1:1,000,000) during their breast reduction.
  Tumescent Solution with dilute epinephrine: Tumescent Solution containing dilute epinephrine (1:1,000,000) only
- Tumescent Solution With Dilute Lidocaine and Epinephrine: Participants in this arm of the study will receive tumescent solution containing both dilute lidocaine (0.05%) and dilute epinephrine (1:1,000,000).
  Tumescent solution with dilute lidocaine and epinephrine: Tumescent Solution containing both dilute lidocaine (0.05%) and dilute epinephrine (1:1,000,000)
Period: Overall Study
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 42 [22 to 70] | 41 [20 to 68] | 41.5 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Mean Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 31 [18 to 55] | 33 [25 to 46] | 32 [18 to 55]
Active Smoker [Number; unit: percentage of participants] | 5 | 15 | 10
History of post-op nausea [Number; unit: percentage of participants] | 20 | 10 | 15
History of previous breast surgery [Number; unit: percentage of participants] | 0 | 25 | 12.5

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Aim 1 is to determine the effect of dilute lidocaine in tumescent solution on post-operative pain following breast reduction surgery. The data points that will be statistically compared will be pain scores determined via a validated pain survey (pain levels on a scale of 0-10 where 10 is the worst pain) and the amount of narcotic medication administered (in Postanesthesia Care Unit (PACU), phase 2 and up to 24 hours post-op) determined from responses to survey questions and by reviewing the medical record.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
score on a scale
  End of PACU Mean Pain Level | 5.47 [0 to 10] | 4.47 [1 to 10]
  First 24 hrs Post-op Mean Current Pain | 4.00 [0 to 9] | 4.28 [1 to 9]
  First 24 hrs Post-op Mean Worst Pain | 6.44 [2 to 10] | 6.68 [2 to 10]
  First 24 hrs Post-op Mean Least Pain | 2.00 [0 to 4] | 2.53 [0 to 9]
Statistical Analysis 1: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; End of PACU Mean Pain Level p-value between arms; Test type: Other; p = 0.24, ANOVA
Statistical Analysis 2: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; First 24 hrs Post-op Mean Current Pain p-value between arms; Test type: Other; p = 0.76, ANOVA
Statistical Analysis 3: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; First 24 hrs Post-op Mean Worst Pain p-value between arms; Test type: Other; p = 0.78, ANOVA
Statistical Analysis 4: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; First 24 hrs Post-op Mean Least Pain p-value between arms; Test type: Other; p = 0.41, ANOVA

2. Primary Outcome: Amount of Post-Operative Narcotic Medication Administered
Description: Aim 1 is to determine the effect of dilute lidocaine in tumescent solution on post-operative pain following breast reduction surgery. The amount of narcotic medication administered (in Postanesthesia Care Unit (PACU), phase 2 and up to 24 hours post-op) determined by reviewing the medical record.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Full Range); unit: mg
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
mg
  PACU IV hydromorphone | 0.89 [0 to 2.4] | 0.55 [0 to 2]
  First 24 hr Post-op oxycodone | 32.19 [0 to 65] | 29.47 [0 to 80]
Statistical Analysis 1: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; PACU IV hydromorphone p-value between arms; Test type: Other; p = 0.10, ANOVA
Statistical Analysis 2: Comparison: Tumescent Solution With Dilute Epinephrine vs Tumescent Solution With Dilute Lidocaine and Epinephrine; First 24 hr Post-op oxycodone p-value between arms; Test type: Other; p = 0.71, ANOVA

3. Secondary Outcome: Post Operative Nausea and Vomiting
Description: The secondary outcomes that will be measured in this study include number of episodes of post-operative nausea (subjective feeling vs. emesis). This data will be attained by reviewing the medical record and through the validated survey questions.
Time Frame: Up to 24 hours following surgery
Measure: Number; unit: episodes
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
episodes
  Nausea | 8 | 10
  Vomiting | 2 | 4

4. Secondary Outcome: Anti-emetic / Intraoperative Medication Administered (mg)
Description: The secondary outcomes that will be measured in this study include the amount of anti-emetic medication used in the first 24 hours post-op. This data will be attained by reviewing the medical record and through the validated survey questions.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Full Range); unit: mg
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
mg
  Mean Intraoperative hydromorphone | 0.98 [0.3 to 1.5] | 1.06 [0 to 2]
  Mean Intraoperative midazolam | 2.00 [2 to 2] | 1.90 [0 to 4]
  Mean Intraoperative ketorolac | 11.25 [0 to 30] | 16.50 [0 to 30]
  Mean Intraoperative dexamethasone | 6.40 [4 to 10] | 6.00 [0 to 10]
  Mean Intraoperative ondansetron | 3.60 [0 to 4] | 4.05 [4 to 5]

5. Secondary Outcome: Anti-emetic / Intraoperative Fentanyl Administered (Measured in Micrograms)
Description: as for outcome 4
Time Frame: Up to 24 hours following surgery
Measure: Mean (Full Range); unit: micrograms
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
micrograms | 131.30 [50 to 300] | 120.00 [0 to 200]

6. Secondary Outcome: Time to Discharge
Description: The patient's medical record will be reviewed to determine the time it took for the patient to be transitioned from the PACU (post anesthesia care unit) till discharge. This includes the time spent in the PACU, time spent in phase 2 and the total time to discharge.
Time Frame: Up to 24 hours following surgery
Population: Time to discharge data not was reported for all participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 14 | 13
minutes | 158 (40.5) | 153 (29.9)

7. Secondary Outcome: Unplanned Hospital Readmission
Description: The patient's medical record will be reviewed to see if the patient was readmitted to the hospital (unplanned) due to complications related to this surgery.
Time Frame: Up to 1 week following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 hr post-op
Arm/Group | Tumescent Solution With Dilute Epinephrine | Tumescent Solution With Dilute Lidocaine and Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tumescent Solution With Dilute Epinephrine (N=20) | Tumescent Solution With Dilute Lidocaine and Epinephrine (N=20)
Nausea (Gastrointestinal disorders) | 8 | 10
Vomiting (Gastrointestinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes